CLINICAL TRIAL: NCT06363903
Title: Autoimmume/Inflammatory Syndrome Induced by Adjuvants (ASIA Syndrome) Caused by Polypropylene Mesh Implantation - a Pilot Study for Diagnostics and Treatment
Brief Title: ASIA-Mesh: a Pilot Study for Diagnostics and Treatment on ASIA Syndrome Caused by Polypropylene Mesh Implantation
Status: Recruiting | Type: Observational
Sponsor: Maxima Medical Center (Other)
Collaborators: Amsterdam UMC (Other); Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Willem A.R. Zwaans, Principal Investigator, Surgeon, Maxima Medical Center
Other Study IDs: 2022-MMC-051
Record Dates: First submitted 2024-02-26; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Autoimmunity; Inguinal Hernia; Stress Urinary Incontinence; Pelvic Organ Prolapse; Implant Complication; Systemic Autoimmune Disease
Keywords: ASIA; Polypropylene; Mesh reaction; Implant; Pilot
MeSH Terms: conditions — Autoimmune Diseases; Hernia, Inguinal; Urinary Incontinence, Stress; Pelvic Organ Prolapse | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood tests, mesh allergy tests, in case of mesh removal: histopathologically prepared explant of mesh
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Included patients: Patients included with index operation that are referred to a participating outpatient clinic and who present with ASIA Syndrome-like complaints occurring after PP implant placement.
  Interventions: Diagnostic Test: mesh allergy test; Diagnostic Test: blood tests; Procedure: Mesh removal

INTERVENTIONS:
Diagnostic Test: mesh allergy test — a 5 mm^2 part of polypropylene mesh will be dissolved in 1 mL Methyl ethyl ketone (MEK), 25 microliters of this solution will be topically applied in a Finn chamber, and a reaction to the topical applicant will be assessed within 48 hours after application.
Diagnostic Test: blood tests — Blood tests for diagnosis of autoimmune diseases will be performed
Procedure: Mesh removal — If wish for mesh removal persists, this procedure can be performed after separate informed consent (within the study), as standard practice of care.

SUMMARY:
In the present pilot study, a possible relation between the implantation of PP mesh for inguinal hernia, vaginal prolapse and SUI repair and subsequent systemic auto-immune complaints is investigated by testing immunologic and allergic responses in fifty patients with suspected ASIA syndrome. Additional value of MAT is investigated and effectiveness of (partial) PP mesh removal for these complaints is assessed. If so, a profound insight in diagnostics and treatment for systematic complaints will be attained that may provide opportunities for future diagnostics.

DETAILED DESCRIPTION:
Worldwide there is a lot of commotion about the effects and complications of various implants. In analogy to patients with silicone breast implants, some patients report various systemic complaints following inguinal polypropylene (PP) mesh implantation, suggesting 'Autoinflammatory/Autoimmunity Syndrome Induced by Adjuvants' (ASIA; Shoenfeld's syndrome) or some other suspected systemic auto-immune/inflammatory response. Although an evidence-based and causal relationship is lacking, patients report serious complaints. Therefore, the investigators recently started seeing these patients at the outpatient clinic and developed a diagnostic workup, including an elaborate anamnesis, conventional immunologic analyses and mesh allergy testing (MAT). Further, in case the implant is removed as part of the treatment due to a persistent wish of the patient, the PP explant will be histologically examined to find additional cues for an auto-immune/inflammatory response (and thus ASIA). So far, evidence on the optimal diagnostic workup for patients with suspected ASIA syndrome is lacking completely.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age and written informed consent obtained;
* Suspected ASIA syndrome after elective hernia, pelvic organ prolapse (POP) surgery, or stress urinary incontinence (SUI) repair, defined as three major ASIA criteria (Table 1), of which the exposure to an external stimulus (PP mesh) is one;
* ASIA complaints evolved after the implantation of PP mesh and were not present before the surgical repair.

Exclusion Criteria:

* Known auto-immune disorders;
* Known malignancies;
* (Low grade) infections or other inflammatory diseases at time of surgery;
* Cognitively impaired individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected auto-immune/inflammatory response or ASIA syndrome will be recruited to one of the outpatient clinics that accept patients with ASIA syndrome complaints. Only referrals will be accepted and no active recruitment will be undertaken.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Positive diagnostic tests | At inclusion. There is no need to repeat this test after first result.
  Rate of positive diagnostic tests of either blood draws or MAT as an indication for presence of an autoimmune disease.

SECONDARY OUTCOMES:
Autoimmune complaints and objective findings in immunologic blood test | At inclusion, questionnaires repeated after 6 and 12 months. Blood tests will not be repeated after tests at inclusion.
  Association between subjective outcomes of autoimmune/inflammatory symptoms and objective findings in blood tests that indicate presence of inflammation or autoimmunity.
Autoimmune complaints and objective findings in mesh allergy test (MAT) | At inclusion, questionnaires repeated after 6 and 12 months. MAT will not be repeated after test at inclusion due to either a positive test (and therefore emergence of immune memory cells) or negative test (and therefore no immune response to mesh at t0)
  Association between subjective outcomes of autoimmune/inflammatory symptoms and objective findings of the mesh allergy test (MAT) that either indicate presence of intolerance to mesh, or indicate no dermal/allergic reaction to the material of the mesh.
Mesh removal and subjective complaints | Follow-up 1 year after surgery. At inclusion, questionnaires repeated after 6 and 12 months.
  Success rate of mesh removal for the resolution of subjective complaints using Tissue Connective Disease Screening Questionnaire (CSQ) and Patient Global Impression of Improvement (PGI-I) questionnaire and ASIA symptoms.
Mesh histopathology | Directly after surgery if surgical mesh removal is deemed safe by the surgeon and preferred by the patient. As attempts will be made to completely remove the mesh, mesh histopathology will only be performed once.
  All explanted meshes will be examined histopathologically to check for granulomatous inflammatory or acute inflammatory reactions surrounding the explant.
Patient demographics | At the start of the inclusion period demographics will be recorded. Demographics will also be recorded for the population undergoing surgery, in combination with Outcome measure 3 of subjective complaints.
  Baseline patient demographics will be collected for all included patients, as well as for patients undergoing surgical mesh removal. Descriptive analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Willem AR Zwaans, MD PhD, Principal Investigator — Maxima Medical Center; Maurits JC Gielen, MD, Study Director — Maxima Medical Center
Locations (3):
- Netherlands (3):
  - Maastricht University Medical Centre, Maastricht, Limburg
  - Maxima Medical Centre, Veldhoven, North Brabant
  - Amsterdam UMC, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Denman MA, Gregory WT, Boyles SH, Smith V, Edwards SR, Clark AL. Reoperation 10 years after surgically managed pelvic organ prolapse and urinary incontinence. Am J Obstet Gynecol. 2008 May;198(5):555.e1-5. doi: 10.1016/j.ajog.2008.01.051. Epub 2008 Mar 20. PMID 18355779
- [Background] Lowenstein E, Moller LA, Laigaard J, Gimbel H. Reoperation for pelvic organ prolapse: a Danish cohort study with 15-20 years' follow-up. Int Urogynecol J. 2018 Jan;29(1):119-124. doi: 10.1007/s00192-017-3395-3. Epub 2017 Jul 3. PMID 28674735
- [Background] Chughtai B, Sedrakyan A, Mao J, Eilber KS, Anger JT, Clemens JQ. Is vaginal mesh a stimulus of autoimmune disease? Am J Obstet Gynecol. 2017 May;216(5):495.e1-495.e7. doi: 10.1016/j.ajog.2016.12.021. Epub 2016 Dec 26. PMID 28034649
- [Background] Chughtai B, Thomas D, Mao J, Eilber K, Anger J, Clemens JQ, Sedrakyan A. Hernia repair with polypropylene mesh is not associated with an increased risk of autoimmune disease in adult men. Hernia. 2017 Aug;21(4):637-642. doi: 10.1007/s10029-017-1591-1. Epub 2017 Feb 23. PMID 28233069
- [Background] Kowalik CR, Zwolsman SE, Malekzadeh A, Roumen RMH, Zwaans WAR, Roovers JWPR. Are polypropylene mesh implants associated with systemic autoimmune inflammatory syndromes? A systematic review. Hernia. 2022 Apr;26(2):401-410. doi: 10.1007/s10029-021-02553-y. Epub 2022 Jan 12. PMID 35020091
- [Background] Cohen Tervaert JW. Autoinflammatory/autoimmunity syndrome induced by adjuvants (Shoenfeld's syndrome) in patients after a polypropylene mesh implantation. Best Pract Res Clin Rheumatol. 2018 Aug;32(4):511-520. doi: 10.1016/j.berh.2019.01.003. Epub 2019 Mar 1. PMID 31174820
- [Background] Muller P, Gurol-Urganci I, Thakar R, Ehrenstein MR, Van Der Meulen J, Jha S. Impact of a mid-urethral synthetic mesh sling on long-term risk of systemic conditions in women with stress urinary incontinence: a national cohort study. BJOG. 2022 Mar;129(4):664-670. doi: 10.1111/1471-0528.16917. Epub 2021 Oct 5. PMID 34524725
- [Background] Zwaans WA, Perquin CW, Loos MJ, Roumen RM, Scheltinga MR. Mesh Removal and Selective Neurectomy for Persistent Groin Pain Following Lichtenstein Repair. World J Surg. 2017 Mar;41(3):701-712. doi: 10.1007/s00268-016-3780-y. PMID 27815571
- [Background] Slooter GD, Zwaans WAR, Perquin CW, Roumen RMH, Scheltinga MRM. Laparoscopic mesh removal for otherwise intractable inguinal pain following endoscopic hernia repair is feasible, safe and may be effective in selected patients. Surg Endosc. 2018 Mar;32(3):1613-1619. doi: 10.1007/s00464-017-5824-2. Epub 2017 Aug 24. PMID 28840390